CLINICAL TRIAL: NCT03848429
Title: Mechanical Complications of Acute Myocardial Infarction: an International Multicenter Cohort Study (CAUTION Study 1)
Brief Title: Mechanical Complications of Acute Myocardial Infarction
Acronym: CAUTION
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL69173.068.19
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Post-Infarction Heart Rupture; Post-Infarction Ventricular Septal Defect; Post-Infarction Mitral Papillary Muscle Rupture
MeSH Terms: conditions — Heart Rupture, Post-Infarction | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery for mechanical complications of acute myocardial infarction — Surgical treatment of post-AMI left ventricular free-wall rupture: sutured and sutureless repair. Surgical treatment of post-AMI ventricular septal defect: infarctectomy and infarct exclusion repair. Surgical treatment of post-AMI papillary muscle rupture: mitral valve repair and replacement

SUMMARY:
Although the incidence of post-AMI mechanical complications has decreased in the last decades, mortality in patients who develop these complications after AMI still remains very high.

Because of the rarity of these post-AMI mechanical complications, the optimal evidence-based therapeutic strategies remain controversial, and little is know on the early clinical results and late follow-up.

Owing to the paucity and limitation of available data, investigations and analysis are required to help clinicians make an early diagnosis of these devastating complications, and offer to patients the appropriate treatment.

"Mechanical complications of acute myocardial infarction: an international multicenter cohort study" (Caution Study 1) is a retrospective, international multicenter clinical trial aimed at evaluating the survival, postoperative outcome and quality of life of patients underwent cardiac surgery for post-AMI mechanical complications.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a major cause of mortality and morbidity worldwide. In the United States cardiovascular disease is the leading cause of death in people older than 65 years. In the current era, a complete recovery after an acute myocardial infarction (AMI) has become the norm. Unfortunately, however, the mortality for some patients remains high. In particular, patients with cardiogenic shock after an AMI have less than a 50% chance of surviving their hospital stay.

Cardiogenic shock in AMI may result from ventricular dysfunction or it may result from mechanical complications requiring emergency surgical treatment; these include: papillary muscle rupture, ventricular free wall rupture and ventricular septal defect.

With the advent of percutaneous coronary intervention (PCI), there has been a significant drop in the incidence of post-infarction mechanical complications.The incidence of mechanical complications after acute ST elevation MI (STEMI) in the APEX-MI trial, where primary PCI was the reperfusion strategy, was 0.9%.

Although the incidence has decreased in the last decades, mortality in patients who develop these complications after AMI still remains very high. Mechanical complications must be carefully searched for in any patient with an acute coronary syndrome and signs of cardiogenic shock. The diagnosis, or even the suspicion, requires urgent surgical referral and in most cases necessitates emergency surgery.

The management of patients with postinfarction mechanical complications requires the consideration of several factors: (i) the extremely poor prognosis without surgical treatment; (ii) the higher mortality risk associated with emergency surgery; (iii) the potential rapid deterioration of initially stable patients.

Data from the Society of Thoracic Surgeons National Database demonstrated an average 43% in-hospital/30-day mortality for surgical treatment of ventricular septal defect. Reports on outcomes in large free wall rupture and papillary muscle rupture cohorts are scarce; based on available data, in-hospital mortality after surgery is around 20-25% for acute mitral regurgitation and 12-36% for ventricular free wall rupture.

In conclusion, because of the rarity of these post-AMI mechanical complications, the optimal evidence-based therapeutic strategies remain controversial, and little is know on the early clinical results and late follow-up.

Owing to the paucity and limitation of available data, investigations and analysis are required to help clinicians make an early diagnosis of these devastating complications, and offer to patients the appropriate surgical treatment. "Mechanical complications of acute myocardial infarction: an international multicenter cohort study" (Caution Study 1) is a retrospective, international multicenter clinical trial aimed at evaluating the survival, postoperative outcome and quality of life of patients underwent cardiac surgery for post-infarction mechanical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old;
* Patients who received surgical treatment for mechanical complications of AMI from January 2001 to December 2018.

Exclusion Criteria:

* Patients who underwent medical/conservative management for post-AMI mechanical complications or cardiac surgery procedures (for example: left ventricular free wall rupture repair) not related with post-AMI complications (for example: traumatic ventricular wall rupture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (≥ 18 years) that required cardiac surgery for mechanical complications of AMI in the participating center from January 2001 to December 2018. Expected population number: 300 patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital survival | Time interval from cardiac surgery to hospital discharge (expected: up to 4 weeks)
  To assess the in-hospital survival rate of patients underwent cardiac surgery for mechanical complications of AMI
Left ventricular free-wall (LVFW) re-rupture | Time interval from cardiac surgery to hospital discharge (expected: up to 4 weeks)
  To assess the LVFWR re-rupture rate of patients underwent post-infarction left ventricular free-wall rupture repair. The presence of LVFW re-rupture will be assessed by echocardiography, or intra-operatively during reoperation.
Ventricular septal defect (VSD) recurrence | Time interval from cardiac surgery to hospital discharge (expected: up to 4 weeks)
  To assess the VSD recurrence rate of patients underwent post-infarction ventricular septal defect repair. The presence of VSD recurrence will be assessed by echocardiography.

SECONDARY OUTCOMES:
Long-term survival | Time interval from hospital discharge to follow-up (expected: up to 100 months)
  To assess the long-term survival rate of patients underwent cardiac surgery for mechanical complications of AMI
Post-operative quality of life | Time interval from hospital discharge to follow-up (expected: up to 100 months)
  To assess the quality of life at follow-up of patients underwent cardiac surgery for mechanical complications of AMI. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems: Level 1: indicating no problem; Level 2: indicating slight problems; Level 3: indicating moderate problems; Level 4: indicating severe problems; Level 5: indicating extreme problems. Higher scores indicate higher levels of health. An unique health state is defined by combining 1 level from each of the 5 dimensions. A total of 3125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code. For example state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Matteucci Matteo, Maastricht, Netherlands

REFERENCES:
- [Result] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Result] Lang IM, Forman SA, Maggioni AP, Ruzyllo W, Renkin J, Vozzi C, Steg PG, Hernandez-Garcia JM, Zmudka K, Jimenez-Navarro M, Sopko G, Lamas GA, Hochman JS. Causes of death in early MI survivors with persistent infarct artery occlusion: results from the Occluded Artery Trial (OAT). EuroIntervention. 2009 Nov;5(5):610-8. doi: 10.4244/eijv5i5a98. PMID 20142183
- [Result] French JK, Hellkamp AS, Armstrong PW, Cohen E, Kleiman NS, O'Connor CM, Holmes DR, Hochman JS, Granger CB, Mahaffey KW. Mechanical complications after percutaneous coronary intervention in ST-elevation myocardial infarction (from APEX-AMI). Am J Cardiol. 2010 Jan 1;105(1):59-63. doi: 10.1016/j.amjcard.2009.08.653. PMID 20102891
- [Result] Rogers WJ, Frederick PD, Stoehr E, Canto JG, Ornato JP, Gibson CM, Pollack CV Jr, Gore JM, Chandra-Strobos N, Peterson ED, French WJ. Trends in presenting characteristics and hospital mortality among patients with ST elevation and non-ST elevation myocardial infarction in the National Registry of Myocardial Infarction from 1990 to 2006. Am Heart J. 2008 Dec;156(6):1026-34. doi: 10.1016/j.ahj.2008.07.030. Epub 2008 Nov 1. PMID 19032996
- [Result] Insam C, Paccaud F, Marques-Vidal P. Trends in hospital discharges, management and in-hospital mortality from acute myocardial infarction in Switzerland between 1998 and 2008. BMC Public Health. 2013 Mar 25;13:270. doi: 10.1186/1471-2458-13-270. PMID 23530470
- [Result] Jennings SM, Bennett K, Lonergan M, Shelley E. Trends in hospitalisation for acute myocardial infarction in Ireland, 1997-2008. Heart. 2012 Sep;98(17):1285-9. doi: 10.1136/heartjnl-2012-301822. Epub 2012 Jul 16. PMID 22802000
- [Result] Arnaoutakis GJ, Zhao Y, George TJ, Sciortino CM, McCarthy PM, Conte JV. Surgical repair of ventricular septal defect after myocardial infarction: outcomes from the Society of Thoracic Surgeons National Database. Ann Thorac Surg. 2012 Aug;94(2):436-43; discussion 443-4. doi: 10.1016/j.athoracsur.2012.04.020. Epub 2012 May 23. PMID 22626761
- [Result] Chevalier P, Burri H, Fahrat F, Cucherat M, Jegaden O, Obadia JF, Kirkorian G, Touboul P. Perioperative outcome and long-term survival of surgery for acute post-infarction mitral regurgitation. Eur J Cardiothorac Surg. 2004 Aug;26(2):330-5. doi: 10.1016/j.ejcts.2004.04.027. PMID 15296892
- [Result] Haddadin S, Milano AD, Faggian G, Morjan M, Patelli F, Golia G, Franchi P, Mazzucco A. Surgical treatment of postinfarction left ventricular free wall rupture. J Card Surg. 2009 Nov-Dec;24(6):624-31. doi: 10.1111/j.1540-8191.2009.00896.x. PMID 20078707
- [Derived] Massimi G, Matteucci M, De Bonis M, Kowalewski M, Formica F, Russo CF, Sponga S, Vendramin I, Colli A, Falcetta G, Trumello C, Carrozzini M, Fischlein T, Troise G, Dato GA, D'Alessandro S, Sardari Nia P, Lodo V, Villa E, Shah SH, Scrofani R, Binaco I, Kalisnik JM, Dell'Uomo M, Pettinari M, Thielmann M, Meyns B, Khouqeer FA, Fino C, Simon C, Musazzi A, Kowalowka A, Deja MA, Pisani A, Batko J, Borghetti V, Ronco D, Di Mauro M, Lorusso R. Repair Versus Replacement in Mitral Valve Papillary Muscle Rupture: A Multicenter Study. Eur J Cardiothorac Surg. 2025 Sep 2;67(9):ezaf284. doi: 10.1093/ejcts/ezaf284. PMID 40845148
- [Derived] Massimi G, Ronco D, De Bonis M, Kowalewski M, Formica F, Russo CF, Sponga S, Vendramin I, Falcetta G, Fischlein T, Troise G, Trumello C, Actis Dato G, Carrozzini M, Shah SH, Coco VL, Villa E, Scrofani R, Torchio F, Antona C, Kalisnik JM, D'Alessandro S, Pettinari M, Sardari Nia P, Lodo V, Colli A, Ruhparwar A, Thielmann M, Meyns B, Khouqeer FA, Fino C, Simon C, Kowalowka A, Deja MA, Beghi C, Matteucci M, Lorusso R. Surgical treatment for post-infarction papillary muscle rupture: a multicentre study. Eur J Cardiothorac Surg. 2022 Jan 24;61(2):469-476. doi: 10.1093/ejcts/ezab469. PMID 34718501